CLINICAL TRIAL: NCT04473794
Title: Diagnostic Strategies, Risk Assessment and Progression of Pancreatic Cysts
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00249790
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Neoplasms; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Surgical Tissue Pancreatic cyst fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study are to determine the natural history of pancreatic cysts and to propose and prospectively validate a diagnostic approach and model for prediction of mucinous versus non-mucinous, and malignant versus non-malignant, pancreatic cysts using a combination of clinical, radiologic, and biomarker characteristics.

DETAILED DESCRIPTION:
Pancreatic cysts are increasingly recognized as incidental lesions due to the widespread use of cross-sectional imaging techniques such as CT and MRI. Twenty percent of all pancreatic cysts are non-inflammatory cystic neoplasms, many of which are mucinous, and therefore have a significant potential for malignant transformation. The primary challenge facing clinicians is the inability of current standard diagnostic tests, including imaging and standard laboratory data, to accurately and reliably discriminate neoplastic from non-neoplastic, and benign from malignant cysts, particularly in patients without symptoms. Therefore, some patients with benign cysts undergo unnecessary costly surveillance and possible avoidable surgical resections, which is associated with high cost, significant morbidity and mortality, while some may not be as aggressively followed. The International Association of Pancreatology (IAP) has published guidelines on the management of the two main types of mucinous cystic lesions: intraductal papillary mucinous neoplasms (IPMNs) and mucinous cystic neoplasms (MCNs). (1) Although these guidelines emphasize the frequency of surveillance and outline the indications for resection, these guidelines have not yet been validated, and these guidelines presume the diagnosis of a mucinous neoplastic cyst has been confirmed prior to surgery. It is unlikely that guidelines that only use clinical and imaging will be able to accurately differentiate benign cysts from those that are pre-malignant or currently harbor malignancy. Hence, there is a critical need for a diagnostic model that more accurately diagnoses neoplastic mucinous and malignant pancreatic cysts as this will improve the management of many patients with pancreatic cysts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years and older
* Referred for assessment of a pancreatic cyst.

Exclusion Criteria:

* Medically ill patients with American Society of Anesthesiologists class 4 or greater.
* Inability to provide informed consent.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of standard care, patients will have a consultation (clinic) visit with a gastroenterologist or surgeon. Patients will be followed per the standard of care at each institution. There are no required study visits. There will be no blinding performed in this study. All patients will receive standard (routine) medical care. No placebo or non-treatment group will be enrolled. There is no treatment failure. Patients will only be removed from the study if patients request this. When the study ends, or if a patient ends his or her participation prematurely, all patients will continue to receive medical and/or surgical care from patients' respective physicians based on currently available published data and clinical experience.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2035-11-01 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical utility of Compcyst in pancreatic cysts as assessed by patient chart review | 15 years
  Compcyst is part of the new standard of care diagnosis of precancerous and benign cystic lesions. Patient charts will be reviewed for clinical, radiological, surgical and pathologic information (all combined into a composite) that will be used to determine if Compcyst as part of the new standard of care is better than the diagnostic measure in the old standard of care in detecting precancerous and benign cystic lesions. Patient records over a 15-year period will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Afghani, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States